CLINICAL TRIAL: NCT06963476
Title: rTMS as Add on Treatment for Substance Use Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Steele 042225; HHC-2025-0073 (Other: Hartford Health Care)
Record Dates: First submitted 2025-05-06; First posted 2025-05-09 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Individuals receiving treatment from Hartford Health Care (HHC) for AUD or OUD will be recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AUD (Experimental): Individuals receiving treatment from HHC for AUD. Participants will be asked to complete a battery of tasks at the prior to the first rTMS session and after the last rTMS session. Each rTMS eligible participant will be scheduled for 5 rTMS visits (to be completed within 2 weeks from start to finish). Each rTMS session will start with finding motor hotspot, the rTMS dose, then application of rTMS. Within AUD participants, random assignment of rTMS site (cTBS at mPFC vs iTBS at l-dlPFC) will occur in sets of 6 thus increasing rTMS site distribution even if a small sample is collected.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS) for AUD
- OUD (Experimental): Individuals receiving treatment from HHC for OUD. Participants will be asked to complete a battery of tasks at the prior to the first rTMS session and after the last rTMS session. Each rTMS eligible participant will be scheduled for 5 rTMS visits (to be completed within 2 weeks from start to finish). Each rTMS session will start with finding motor hotspot, the rTMS dose, then application of rTMS. Within OUD participants, random assignment of rTMS type (cTBS vs iTBS ) applied to l-dlPFC will occur in sets of 6 thus increasing rTMS site distribution even if a small sample is collected.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS) for OUD

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) for AUD — Transcranial magnetic stimulation (TMS) is a noninvasive form of brain stimulation in which a changing magnetic field is used to cause electric current at a specific area of the brain through electromagnetic induction. To administer TMS, a stimulator equipped with a figure-8 coil will be used. Two separate coils will be used that are similar in appearance and acoustic properties. One active, unblinded, coil will be used to determine resting motor threshold (RMT) and deliver pulses for the recruitment curves; the other coil will be used to deliver rTMS. rTMS stimulation will be targeted using standard EEG electrode locations: FP1 for mPFC and F3 for l-dlPFC.
  Arms: AUD
Device: repetitive transcranial magnetic stimulation (rTMS) for OUD — Description: Transcranial magnetic stimulation (TMS) is a noninvasive form of brain stimulation in which a changing magnetic field is used to cause electric current at a specific area of the brain through electromagnetic induction. To administer TMS, a stimulator equipped with a figure-8 coil will be used. Two separate coils will be used that are similar in appearance and acoustic properties. One active, unblinded, coil will be used to determine resting motor threshold (RMT) and deliver pulses for the recruitment curves; the other coil will be used to deliver rTMS. rTMS stimulation will be targeted using standard EEG electrode location F3 for l-dlPFC.
  Arms: OUD

SUMMARY:
This pilot study is designed to test feasibility and superiority of rTMS types and target locations for the optimal rTMS intervention for individuals seeking treatment for Alcohol Use Disorder (AUD) or Opioid Use Disorder (OUD).

The critical questions this study seeks to answer are: which rTMS type applied to l-dlPFC in OUD participants will induce the greatest reduction of opioid use post-treatment? Is inhibitory rTMS applied to medial prefrontal cortex (mPFC) more effective than excitatory rTMS applied to l-dlPFC at reducing alcohol use post treatment in AUD participants?

DETAILED DESCRIPTION:
Aim 1: To assess feasibility of applying rTMS within a residential treatment center. Feasibility will be assessed by 1) recruitment of sufficient numbers of AUD and OUD participants; 2) completion of the rTMS intervention; 3) retention of follow-up at the 4-week interval.

Aim 2: To assess superiority of mPFC cTBS compared to l-dlPFC iTBS to reduce alcohol use in AUD patients post-treatment. Superiority will be assessed by evaluating 1) treatment engagement at the 4-week interval (e.g., number of prescribed AUD treatments addended); 2) reduction of drinks/day post-treatment, compared to pre-treatment; 3) reduction of heavy drinking days (e.g., >5 drinks/day) post-treatment, compared to pre-treatment.

Aim 3: To assess superiority of l-dlPFC iTBS to l-dlPFC cTBS to reduce opioid use in OUD patients post-treatment. Superiority will be assessed by evaluating 1) treatment engagement at the 4-week interval (e.g., number of prescribed OUD treatments addended); 2) reduction of opioids used post-treatment, compared to pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give valid informed consent in English.
* Absence of cognitive impairment: IQ equivalent of ≥ 70 on the WRAT.
* Receiving treatment for either AUD or OUD

Exclusion Criteria:

* History of any neurological disorder that would increase seizure risk from rTMS such as stroke, brain lesions, previous neurosurgery, any history of seizure or fainting episode of unknown cause, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than one month.
* Current meeting withdrawal criteria for alcohol: AUD participants will not meet for clinically significant alcohol withdrawal: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) ≤ 5.
* First-degree family history of epilepsy or multiple sclerosis.
* Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps or sensors, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object in the body that precludes rTMS administration.
* Current use of anti- or pro-convulsive action.
* Use of benzodiazepines in the last 48 hours prior to rTMS. Benzodiazepines are used during alcohol withdrawal management but then are discontinued prior to recruitment into the study. Therefore, rTMS eligible participants will not continue taking benzodiazepines.
* Lifetime history of schizophrenia, bipolar disorder, mania.
* History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke, or transient ischemic attack.
* Pregnant or lactating women.
* TMS contraindications.
* Treatment center discharge date does not allow for scheduling of all 5 rTMS days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants that successfully complete the study | 4-weeks post-treatment
  Successful completion of the study is defined as completing the rTMS protocol and the 4-week post-treatment follow-up.
Mean number of drinks per day | 4-weeks post-treatment
  A timeline follow-back will be used to assess number of drinks per day.
Mean number of heavy drinking days | 4-weeks post-treatment
  A timeline follow-back will be used to assess number of heavy drinking days.
Opioid use | 4-weeks post-treatment
  A timeline follow-back will be used to assess the quantity of opioids used in bags.

CONTACTS AND LOCATIONS:
Overall Officials: Vaughn R Steele, PhD, Principal Investigator — Yale University
Locations (1):
- Hartford Healthcare, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No